CLINICAL TRIAL: NCT01836367
Title: An Investigator-Initiated Study to Assess the Degree of Irritation After a Second Cycle of Ingenol Mebutate 0.015% Gel in the Treatment of Actinic Keratoses (AK) on the Face and Scalp
Brief Title: Ingenol Mebutate 0.015% Gel in the Treatment of Actinic Keratoses (AK) on the Face and Scalp
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Principal Investigator, Mark Lebwohl, Chairman, Dept of Dermatology, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: GCO 13-0026
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; Face; Scalp; Ingenol Mebutate
MeSH Terms: conditions — Keratosis, Actinic; Facies | interventions — 3-ingenyl angelate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ingenol Mebutate 0.015% (Experimental): two cycles of ingenol mebutate 0.015%
  Interventions: Drug: Ingenol Mebutate 0.015%

INTERVENTIONS:
Drug: Ingenol Mebutate 0.015% — Picato
  Other Names: ingenol mebutate 0.015% qdaily x 3 days for two cycles

SUMMARY:
Actinic keratoses (AK) are common cutaneous lesions associate with chronic ultraviolet radiation exposure. While most authorities consider AK as a pre-malignant lesion, some consider it as an incipient squamous cell carcinoma (SCC). Among the current therapies for the treatment of AK are excisional surgery, cryosurgery, electrodesiccation and curettage, topical chemotherapy and light therapies. Cryosurgery is considered the gold standard for therapy, however as with other lesion-directed therapies, cryosurgery does not treat subclinical lesions in the surrounding skin. Ingenol mebutate is the active compound in the sap from Euphorbia peplus L. (E. peplus). Topical ingenol mebutate treatment has been approved for the treatment of AKs. The goal of AK therapy for all physicians is to provide an effective, tissue-sparing treatment with good cosmetic results. Ingenol mebutate gel 0.015% has shown to not only have a high clearance rate but also a transient localized inflammatory skin response that resolves quickly without sequelae. However, one common fear about ingenol mebutate is that it's mechanism of action is purely destructive to both AKs and healthy skin, and that retreatment would produce an equally, if not more, caustic result on the skin such as severe erosion, scaling, and erythema. It is our hope to debunk this misconception and demonstrate that reapplication of a second cycle of ingenol mebutate would result in lower LSR scores compared to the LSR in the first cycle of application. We plan to treat 20 subjects. Each qualifying subject will have at least 4-8 non-hypertrophic AKs in a 25 cm2 treatment area on the face or scalp. All subjects will be treated with two cycles of ingenol mebutate 0.015%. The first cycle will be started on Day 1, and the second cycle will be started on Day 29 (four weeks apart). Subjects will utilize the once daily for three days regimen for both cycles.

DETAILED DESCRIPTION:
We plan to treat 20 subjects. Each qualifying subject will have at least 4-8 non-hypertrophic AKs in a 25 cm2 treatment area on the face or scalp. All subjects will be treated with two cycles of ingenol mebutate 0.015%. The first cycle will be started on Day 1, and the second cycle will be started on Day 29 (four weeks apart). Subjects will utilize the once daily for three days regimen for both cycles. For the first cycle of study application, subjects will be followed on day 1, day 2, and day 4 during treatment; on day 1 baseline photographs will be taken, on day 2 LSR will be assessed and visual analog scale (VAS) regarding perceived irritation will be conducted, and on day 4 LSR, VAS and photographs will be taken. Post-treatment follow-up will be conducted on day 8 and day 15, in which LSR will be assessed and photographs taken. Approximately four weeks later, a second cycle of once daily for three day regimen of ingenol mebutate 0.015% will be applied to the same treatment area on the face or scalp. Subjects will be followed during treatment on day 29, day 30 and day 32; on day 29 LSR and photographs will be taken, on day 30 LSR will be assessed and VAS conducted, and on day 32 LSR, VAS and photographs will be taken. Post-treatment follow-up for the second cycle of application will occur on day 36, day 43, and day 56. During these post-treatment follow-up visits LSR and photographs will be taken. LSR scores from day 4 and day 32 will be assessed by a blinded observer. Lastly, on day 29 and day 56 the patient's treatment satisfaction will be evaluated on a 10 point visual analog scale (VAS). Consequently, there will be a total of 11 visits during a 56 day period.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years old.
* Subjects must be in good general health as confirmed by the medical history.
* Subjects must be able to read, sign, and understand the informed consent
* Subjects have at least 4-8 clinically typical, visible, non-hypertrophic actinic keratoses on the face or scalp in a 25 cm2 area.
* Subject must be willing to forego any other treatments on the face or scalp, including tanning bed use and excessive sun exposure while in the study.
* Subject is willing and able to participate in the study as an outpatient, making frequent visits to the study center during the treatment and follow-up periods and to comply with all study requirements including concomitant medication and other treatment restrictions.
* If subject is a female of childbearing potential she must have a negative urine pregnancy test result prior to study treatment initiation and must agree to use an approved method of birth control while enrolled in the study.

Exclusion Criteria:

* Subjects with a history of melanoma anywhere on the body.
* The second cycle of ingenol mebutate 0.015% should only be applied if the skin is healed from the first cycle of ingenol mebutate 0.015%.
* Subjects with an unstable medical condition as deemed by the clinical investigator.
* Subjects with non-melanoma skin cancer on the face or scalp.
* Subjects with any dermatologic disease in the treatment area that may be exacerbated by the treatment proposed or that might impair the evaluation of AKs.
* Subjects who have previously been treated with ingenol mebutate: on the face or scalp in the past 6 months; or outside of the study area within the past 30 days.
* Women who are pregnant, lactating, or planning to become pregnant during the study period.
* Subjects who have experienced a clinically important medical event within 90 days of the visit (e.g., stroke, myocardial infarction, etc).
* Subjects who have active chemical dependency or alcoholism as assessed by the investigator.
* Subjects who have known allergies to any excipient in the study gel.
* Subjects who are currently participating in another clinical study or have completed another clinical study with an investigational drug or device on the study area within 30 days prior to study treatment initiation.
* Subjects who have received any of the following within 90 days prior to study treatment initiation:

  * interferon or interferon inducers
  * cytotoxic drugs
  * immunomodulators or immunosuppressive therapies (inhaled/ intranasal steroids are permitted)
  * oral or parenteral corticosteroids
  * topical corticosteroids if greater than 2 gm/day
  * any dermatologic procedures or surgeries on the study area (including any AK treatments)
* Subjects who have used any topical prescription medications on the study area within 30 days prior to study treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Degree of Irritation after two cycles of ingenol mebutate | up to 1 year
  To evaluate the degree of irritation, as measured by local skin reactions (LSR), after a second cycle of ingenol mebutate gel to the face or scalp through photography assessed by a blinded observer.

SECONDARY OUTCOMES:
Degree of Irritation 1 day post application of first and second cycle of ingenol mebutate | up to 1 year
  To evaluate and compare the degree of irritation, as measured by LSR, that occurs one (1) day post-application of the first and second cycle of ingenol mebutate gel to the face or scalp.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lebwohl, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States